CLINICAL TRIAL: NCT00117858
Title: Double Blind Trial of DC Polarization in FTD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050180; 05-N-0180
Record Dates: First submitted 2005-07-07; First posted 2005-07-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-05-10

CONDITIONS: Dementia
Keywords: Frontal Lobe; Language; Behavior; Degenerative Diseases; Pick's Disease; Frontotemporal Dementia; FTP
MeSH Terms: conditions — Dementia; Language; Behavior; Pick Disease of the Brain; Frontotemporal Dementia

INTERVENTIONS:
Procedure: Anodal DC polarization of left prefrontal cortex

SUMMARY:
This project is designed to test how direct current (DC) electrical polarization of the brain affects language and behavior in patients with frontotemporal dementia (FTD). FTD is the second most common form of dementia after Alzheimer's disease. It causes profound disturbances of language and other cognitive functions and often results in highly disruptive behavior. There is no effective treatment for the behavioral disorder or cognitive deficits in FTD. In an earlier study, the researchers used DC polarization to the primary motor cortex to enhance prefrontal function in healthy subjects. The experiment resulted in greater verbal fluency. In a separate study of five patients with FTD, a similar effect on verbal fluency was produced. The object of the current study is to replicate these findings in a larger group of patients and to see if the results carry over into "real world" behavior.

Participants will be 20 patients aged 35 to 75 years with FTD, referred to the Cognitive Neuroscience Section.

Participants will be tested in two sessions, separated by at least 48 hours. In one session they will receive 40 minutes of anodal DC polarization; in the other they will receive 40 minutes of sham polarization. Participants will be tested for language, memory, and reaction time before and 20 minutes after the polarization. For the behavior portion of the study, the Neuropsychiatric Inventory will be completed by an investigator with the caretaker on admission (covering the preceding week) and again, by telephone, 1 week after discharge, to cover the first week home.

Participants will receive no lasting benefit as a result of the study, but the study is likely to yield generalizable knowledge on the effects of DC polarization treatment in FTD.

DETAILED DESCRIPTION:
Introduction: In a recent sham-controlled pilot study we showed that surface anodal DC polarization can improve verbal fluency in patients with frontotemporal dementia (FTD). This study is designed to extend those findings in a double blind trial. Objective: To see whether surface anodal DC polarization can improve verbal fluency and a global measure of behavior in FTD patients. Design: We propose to treat 20 FTD patients anodal and sham DC polarization in a double blind, crossover trial. Outcome Measures: The primary outcome measures are verbal fluency and the score on the Neuropsychiatric Index, a commonly used scale for behavioral problems in dementia. Secondary outcomes will include a modified behavioral scale, administered every 12 hours during the study, a standard neurobehavioral rating scale, some experimental tests of dominant frontal lobe function and a control task that we do not expect to be affected.

ELIGIBILITY:
* INCLUSION CRITERIA

Patients must:

* meet diagnostic criteria for FTD (Knopman et al., 2005)
* be capable of understanding and cooperating with task instructions
* be fluent enough to generate at least three words in one category in one minute
* be between ages 35 to 75
* be right handed.

EXCLUSION CRITERIA

Presence of metal (prostheses, electrodes, other medical hardware, shrapnel) in the cranial cavity

Broken skin in the area of the electrodes

Inability to comprehend the experiment or to cooperate with treatment or testing

Any uncontrolled medical problem

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-06-28; Study Completion 2007-05-10

PRIMARY OUTCOMES:
Verbal fluency and the score on the Neuropsychiatric Index, a commonly used scale for behavioral problems in dementia.

SECONDARY OUTCOMES:
Modified behavioral scale, administered every 12 hours during the study, a standard neurobehavioral rating scale, some experimental tests of dominant frontal lobe function and a control task that we do not expect to be affected.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425